CLINICAL TRIAL: NCT01609361
Title: Benefit of Rehabilitation Program in Colorectal Laparoscopic Surgery
Brief Title: Benefit of Rehabilitation Program in Colorectal Surgery
Acronym: REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P111006; IDRCB (Other: 2011-A00803-38)
Record Dates: First submitted 2012-04-20; First posted 2012-06-01 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Rehabilitation program; Fast track surgery; Laparoscopic colorectal resection; Colorectal cancer; Morbidity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Standard surgery + Standard care (No Intervention): standard surgery and Standard care after surgery
- 2: Laparoscopy + Rehabilitation program (Other): Laparoscopic colorectal surgery with rehabilitation program
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — Rehabilitation program including specific anesthetic drugs, post operative fast track recovery (early diet, mobilisation, antalgics)
  Arms: 2: Laparoscopy + Rehabilitation program

SUMMARY:
Rehabilitation program improves operative results following conventional open colorectal surgery. Very few data are available on such program in laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
The aim is to assess rehabilitation program in laparoscopic colorectal surgery in terms of 30 days peri operative complications

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Colorectal cancer
* Inform and consent form signed
* Patient has valid health insurance/coverage
* Functional capacity ≥ 4 METs (metabolic equivalents) (up 1 floor without stopping, walking down the street 5-7km / h, major domestic activities)
* Patients with laparoscopic resection for colorectal cancer including abdominoperineal resection

Inclusion Criteria (arm : Laparoscopy + Rehabilitation program):

* Tobacco and alcohol weaning

Exclusion Criteria:

* MBI < 18kg/m2
* severe malnutrition
* Metastatic colorectal cancer
* Buzby Index <83
* Combined surgery (hepatic resection or segmental resection of small intestine)
* Urgent surgery
* Pregnancy or maternal breastfeeding
* Body mass index (BMI)> 30 kg/m2
* Abdominoperineal resection
* Subtotal colectomy
* Total proctocolectomy
* Cons to Naropin Xylocaine, droperidol, ketamine
* Patient with a history of peptic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post operative morbidity at 30 days according to DINDO CLAVIEN classification | 30 days
  Post operative morbidity at 30 days according to DINDO CLAVIEN classification (grade I to IV)

SECONDARY OUTCOMES:
Mortality according to DINDO CLAVIEN classification | up to 30 days
  Mortality according to DINDO CLAVIEN classification (grade V)
Hospital stay and readmissions | up to first month
  Initial hospital stay and possible unscheduled readmissions
Intravenous perfusion stay | participants will be followed until the end of hospitalization an expected average of 2 weeks
Global (SF36) quality of life | Preoperative and at 1, 3, 6 months
  Global (SF36) and specific (GIQLI) quality of life Preoperative and at 1, 3, 6 months
Specific (GIQLI) quality of life | Preoperative and at 1, 3, 6 months
  Global (SF36) and specific (GIQLI) quality of life Preoperative and at 1, 3, 6 months
Duration of laxation (gas and stool) | up to hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie Colorectale / Hôpital Beaujon, Clichy, France